CLINICAL TRIAL: NCT00824746
Title: Retreatment of Gefitinib in the Patients With Non-small Cell Lung Cancer (NSCLC) Previously Responded to Gefitinib A Single Arm, Open Label, Phase II Study
Brief Title: Study of Gefitinib Retreatment in Non-Small Cell Lung Cancer (NSCLC)
Acronym: ReGaiN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Young-Chul Kim, Professor, Chonnam National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D791JL00001
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Results first posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Gefitinib; Recurrence; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gefitinib retreatment group (Experimental): Gefitinib retreatment
  Interventions: Drug: Gefitinib retreatment

INTERVENTIONS:
Drug: Gefitinib retreatment — phase II trial of Gefitinib retreatment for the advanced or metastatic (IIIb and IV) NSCLC patients who previously responded to gefitinib And progressive disease should be observed with at least one prior regimen following previous EGFR-TKI failure.
  Other Names: Iressa

SUMMARY:
A single arm, open label, prospective, phase II trial of Gefitinib retreatment for the advanced or metastatic (IIIb and IV) NSCLC patients who previously responded to gefitinib And progressive disease should be observed with at least one prior regimen following previous gefitinib failure.

Primary endpoint

* to assess Disease Control Rate (Remission + Stable disease)

Secondary endpoints

* to assess the progression free survival

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or progressive Non-Small Cell Lung Cancer (NSCLC) stage IV or IIIB patients after chemotherapy following gefitinib failure
* Male and female patients aged over 18 years
* World Health Organization (WHO) performance status 0-2 (those with performance status 2 must have been stable with no deterioration over the previous 2 weeks)
* Had at least stable disease with previous Gefitinib treatment
* Had at least one anticancer agent therapy after gefitinib failure ;Following treatment with another epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKIs)- erlotinib or other TKIs should not be included in anticancer agent therapy.
* The current approved indication of Gefitinib is 2nd or 3rd line monotherapy for recurrent or metastatic NSCLC. However, in practice with off-label indication, it can also be used as a 1st line treatment at the patient's own expenses. Thus, in this trial gefitinib retreatment will be 3rd line or more.
* Measurable lesion according to Response Evaluation Criteria in Solid Tumors(RECIST) with at least one measurable lesion not previously irradiated, unless disease progression has been documented at that site.
* Provision of written informed consent
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Evidence of clinically active Interstitial Lung Diseases (Patients with chronic, stable, radiographic changes who are asymptomatic need not be excluded)
* Expected life expectancy less than 2 months
* Known severe hypersensitivity to gefitinib or any of the excipients of this product
* Any unresolved chronic toxicity greater that Common Terminology Criteria (CTC) grade 2 from previous anticancer therapy
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* Serum bilirubin greater than 3 times the upper limit of reference range (ULRR)
* Aspartate aminotransferase (AST/SGOT) or alanine aminotransferase (ALT/SGPT) ≥ 2.5 x Upper Limit Normal (ULN) if no demonstrable liver metastases (or >5 x in presence of liver metastases)
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study
* Pregnancy or breast-feeding women (women of child¬bearing potential). Women of childbearing potential must practice acceptable methods of birth control to prevent pregnancy.
* Newly diagnosed central nervous system (CNS) metastases that have not yet been treated with surgery and/or radiation. Patients with previously diagnosed and treated CNS metastases or spinal cord compression may be considered if they have evidence of clinically stable disease (no steroid therapy or steroid dose being tapered) for at least 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young-Chul Kim, MD, PhD, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do, South Korea

REFERENCES:
- [Result] Oh IJ, Ban HJ, Kim KS, Kim YC. Retreatment of gefitinib in patients with non-small-cell lung cancer who previously controlled to gefitinib: a single-arm, open-label, phase II study. Lung Cancer. 2012 Jul;77(1):121-7. doi: 10.1016/j.lungcan.2012.01.012. Epub 2012 Feb 12. PMID 22333554

RESULTS

PARTICIPANT FLOW:
Groups:
- Gefitinib Retreatment Group: Gefitinib retreatment group Patients who were previously treated with gefitinib followed by at least one line of cytotoxic chemotherapy can be enrolled to this retreatment group.
Period: Overall Study
Arm/Group | Gefitinib Retreatment Group
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Gefitinib retreatment
Arm/Group | Single Arm
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 64.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 3
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 23

OUTCOME MEASURES:

1. Secondary Outcome: Progression - Free Survival of Patients Retreated With Gefitinib
Description: Progression is defined, using RECIST (V1.1), as a measurable increase in the smallest dimension of any target or non-target lesion, or the appearance of new lesions, since baseline using CT scan every 8 weeks.
Time Frame: two year
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Gefitinib Retreatment Arm: Gefitinib retreatment arm
Arm/Group | Gefitinib Retreatment Arm
Number analyzed (Participants) | 23
days | 103 [70 to 134]

2. Primary Outcome: Disease Control(DC) Rate of Gefitinib Retreatment Per RECIST Criteria (V1.1) and Assessed by CT
Description: Evaluation of treatment response by computed tomography (CT) was performed after the first 4 weeks according to version 1.1 of the guidelines set out by Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Disease control rate (DCR) was defined as the percentage sum of best tumor response of complete response (CR), partial response (PR), and stable disease (SD).
Time Frame: 8 weeks
Population: we analysed the data of 23 patients who were enrolled to this study(intention-to-treat (ITT) population).
Measure: Number (95% Confidence Interval); unit: percentage of participant with DC
Arm/Group | Gefitinib Retreatment Group
Number analyzed (Participants) | 23
percentage of participant with DC | 65.2 [42.7 to 83.6]

3. Secondary Outcome: Overall Survival
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Single Arm
Number analyzed (Participants) | 23
days | 343 [235 to 409]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 3/23
Other Adverse Events (participants affected / at risk) | 10/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=23)
disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=23)
Skin rash (Skin and subcutaneous tissue disorders) | 8 (8)
diarrhea (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Our study has several limitations such as lack of generalizability outside a clinically and molecularly enriched population and the small number of repeat biopsies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less